CLINICAL TRIAL: NCT00201487
Title: Choline Quantification in Breast Cancer by MRS
Status: Withdrawn | Type: Observational
Why Stopped: We chose to use an exsisting NMR pulse sequence already established and available at the hospital.
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Norwegian Women´s Public Health Association (Other)
Responsible Party: Sponsor
Other Study IDs: 11870
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Choline has been found in increased concentration in breast cancer patients. Hypothesis: The choline signal as observed by MRS is sensitive to treatment, and a positive response to treatment will give a reduction in choline concentration.

The purpose of this study is to establish methods for quantification of choline in breast cancer by MRS

DETAILED DESCRIPTION:
1. Establishment of new MRS sequence for choline quantification of choline. This sequence is choline-selective, and signals from water and lipids are suppressed simultaneously.
2. Compare to different methods for choline quantification. The first method is quantification through an external phantom standard, containing a known concentration of choline. The other method is based on the utilisation of internal water signal as a reference.

Both calculations can be performed from the same MR exam. Ten patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer

Exclusion Criteria:

-

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tone Bathen, PhD, Principal Investigator — NTNU, Faculty of medicine,